CLINICAL TRIAL: NCT05877209
Title: Screening of Nutritional Status and Sarcopenia Among Inflammatory Bowel Disease Patients in Assuit University Hospital
Brief Title: Screening of Nutritional Status and Sarcopenia Among Patients With IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Mohamed Refaat Askalany, Doctor / Principal investigator, Assiut University
Other Study IDs: NRS score in IBD
Record Dates: First submitted 2023-04-02; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Screening of malnutrition in patients with IBD and its relation to severity of the disease.
2. Determination of severity of malnutrition in IBD patients.
3. Assessment of Sarcopenia in patients with IBD.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) encompasses Crohn's disease (CD) and ulcerative colitis (UC) is a chronic, relapsing, inflammatory disorder of the digestive tract that characteristically develops in adolescence and early adulthood. IBD is associated with inflammation and negative nutrient balance, which is a risk factor for malnutrition. Multiple definitions of malnutrition have been proposed in literature. The early definitions of malnutrition referred to a state of under nutrition. Subsequently, an imbalance of nutrients, either deficiency or excess, was included in the definition. World Health Organization (WHO) defines malnutrition as deficiency, excess, or imbalance in a person's intake of energy and/or nutrients. The reported prevalence of malnutrition in IBD varies between 16 % and 75%. Several studies have reported a prevalence of weight loss in 70%-80% of hospitalized IBD patients and in 20%-40% of outpatients with CD. Several factors contribute to malnutrition in IBD patients. It is known that a reduced oral food intake is a main determinant of malnutrition in patients with IBD. Several mechanisms are involved in the reduction of food intake. Patients with active IBD often experience loss of appetite due to nausea, vomiting, abdominal pain, and diarrhea. Medications may also induce nausea, vomiting, or anorexia. Glucocorticoids often reduce phosphorus, zinc, and calcium absorption and may lead to osteoporosis. Long-term sulfasalazine therapy, a folic acid antagonist, might be related to anemia. Hospitalization itself or prolonged restrictive diet may lead to a significant reduction of food intake. The severity of malnutrition in IBD patients is dependent on the activity, duration and extent of the disease. In particular, on the magnitude of the inflammatory systemic response mediated by pro-inflammatory cytokines such as tumor necrosis factor-alpha (TNF) and interleukins-1 and -6, which can increase catabolism and lead to anorexia. Sarcopenia has been defined by the European Working Group on Sarcopenia (EWGSOP) combining low muscle strength, low muscle quantity/quality, and low physical performance. There has been a major change from the original operational definition, as low muscle strength was added as a prerequisite to definitions based only on the detection of low muscle mass. In addition, low physical performance is considered a predictor for poor outcomes; thus, such measures are useful to classify the severity of sarcopenia. Nutritional status is traditionally measured with anthropometric tests including height, weight, body mass index (BMI), body circumferences (waist, hip, and limbs), and skinfold thickness. These parameters improve with IBD treatment but may not reflect changes in body composition. The purpose of the NRS-2002 system is to detect the presence of under nutrition and the risk of developing under nutrition in the hospital setting. It contains the nutritional components of Malnutrition Universal Screening Test (MUST). In addition, a grading of severity of disease as a reflection of increased nutritional requirements. With the prototypes for severity of disease given, it is meant to cover all possible patient categories in a hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years old and diagnosed to have IBD (UC or CD). The diagnosis of IBD will be based on clinical, laboratory, radiological, endoscopic and/or histopathological data.
* Naïve IBD patients or those currently on treatment

Exclusion Criteria:

* Patients undergoing intentional weight loss plan.
* Patients with Cardiac Diseases.
* Patients with Liver diseases
* Patients with Thyroid active diseases.
* Pregnant women with IBD.
* Diabetic patients.
* Patients with extra-intestinal malignancies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Screening of malnutrition in patients with IBD using and its relation to severity of the disease. | Baseline
  screening of malnutrition in patients with IBD using Nutritional Risk Screening score

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Kamel, professor, Study Director — Assiut University

REFERENCES:
- [Background] Goh J, O'Morain CA. Review article: nutrition and adult inflammatory bowel disease. Aliment Pharmacol Ther. 2003 Feb;17(3):307-20. doi: 10.1046/j.1365-2036.2003.01482.x. PMID 12562443
- [Background] Donnellan CF, Yann LH, Lal S. Nutritional management of Crohn's disease. Therap Adv Gastroenterol. 2013 May;6(3):231-42. doi: 10.1177/1756283X13477715. PMID 23634187
- [Background] Casanova MJ, Chaparro M, Molina B, Merino O, Batanero R, Duenas-Sadornil C, Robledo P, Garcia-Albert AM, Gomez-Sanchez MB, Calvet X, Trallero MDR, Montoro M, Vazquez I, Charro M, Barragan A, Martinez-Cerezo F, Megias-Rangil I, Huguet JM, Marti-Bonmati E, Calvo M, Campdera M, Munoz-Vicente M, Merchante A, Avila AD, Serrano-Aguayo P, De Francisco R, Hervias D, Bujanda L, Rodriguez GE, Castro-Laria L, Barreiro-de Acosta M, Van Domselaar M, Ramirez de la Piscina P, Santos-Fernandez J, Algaba A, Torra S, Pozzati L, Lopez-Serrano P, Arribas MDR, Rincon ML, Pelaez AC, Castro E, Garcia-Herola A, Santander C, Hernandez-Alonso M, Martin-Noguerol E, Gomez-Lozano M, Monedero T, Villoria A, Figuerola A, Castano-Garcia A, Banales JM, Diaz-Hernandez L, Arguelles-Arias F, Lopez-Diaz J, Perez-Martinez I, Garcia-Talavera N, Nuevo-Siguairo OK, Riestra S, Gisbert JP. Prevalence of Malnutrition and Nutritional Characteristics of Patients With Inflammatory Bowel Disease. J Crohns Colitis. 2017 Dec 4;11(12):1430-1439. doi: 10.1093/ecco-jcc/jjx102. PMID 28981652
- [Background] Unal NG, Oruc N, Tomey O, Omer Ozutemiz A. Malnutrition and sarcopenia are prevalent among inflammatory bowel disease patients with clinical remission. Eur J Gastroenterol Hepatol. 2021 Nov 1;33(11):1367-1375. doi: 10.1097/MEG.0000000000002044. PMID 33470696
- [Background] Lanfranchi GA, Brignola C, Campieri M, Bazzocchi G, Pasquali R, Bassein L, Labo G. Assessment of nutritional status in Crohn's disease in remission or low activity. Hepatogastroenterology. 1984 Jun;31(3):129-32. PMID 6469202
- [Background] Hartman C, Eliakim R, Shamir R. Nutritional status and nutritional therapy in inflammatory bowel diseases. World J Gastroenterol. 2009 Jun 7;15(21):2570-8. doi: 10.3748/wjg.15.2570. PMID 19496185
- [Background] Hanauer SB, Stathopoulos G. Risk-benefit assessment of drugs used in the treatment of inflammatory bowel disease. Drug Saf. 1991 May-Jun;6(3):192-219. doi: 10.2165/00002018-199106030-00005. PMID 1676590
- [Background] Singleton JW, Law DH, Kelley ML Jr, Mekhjian HS, Sturdevant RA. National Cooperative Crohn's Disease Study: adverse reactions to study drugs. Gastroenterology. 1979 Oct;77(4 Pt 2):870-82. PMID 38177
- [Background] Hebuterne X, Filippi J, Al-Jaouni R, Schneider S. Nutritional consequences and nutrition therapy in Crohn's disease. Gastroenterol Clin Biol. 2009 Jun;33 Suppl 3:S235-44. doi: 10.1016/S0399-8320(09)73159-8. PMID 20117347
- [Background] Lucendo AJ, De Rezende LC. Importance of nutrition in inflammatory bowel disease. World J Gastroenterol. 2009 May 7;15(17):2081-8. doi: 10.3748/wjg.15.2081. PMID 19418580
- [Background] Cabre E, Gassull MA. Nutrition in inflammatory bowel disease: impact on disease and therapy. Curr Opin Gastroenterol. 2001 Jul;17(4):342-9. doi: 10.1097/00001574-200107000-00008. PMID 17031181
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Gerasimidis K, McGrogan P, Edwards CA. The aetiology and impact of malnutrition in paediatric inflammatory bowel disease. J Hum Nutr Diet. 2011 Aug;24(4):313-26. doi: 10.1111/j.1365-277X.2011.01171.x. Epub 2011 May 13. PMID 21564345
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673